CLINICAL TRIAL: NCT04055259
Title: Six-Month Randomized Controlled Trial of Text-Based Mobile Health and Wellness Coaching for Weight Loss
Brief Title: A Mobile Health and Wellness Coaching Intervention for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: Auburn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-278 MR 1707
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Overweight and Obesity; Health Behavior
Keywords: Health and Wellness Coaching
MeSH Terms: conditions — Overweight; Obesity; Health Behavior | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile Health and Wellness Coaching (Experimental)
  Interventions: Behavioral: mobile Health and Wellness Coaching
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: mobile Health and Wellness Coaching — Participants in the mobile health and wellness coaching (mHWC) group received text-based mHWC messages and did not return to the clinic until the end of the 6 month intervention. Messages were sent at least weekly and focused on facilitating the adoption and maintenance of health behaviors related to diet, physical activity and sleep to promote weight loss. Participants could respond via text at any time. The Nudge platform was used for all messaging.
  Arms: mobile Health and Wellness Coaching
Behavioral: Usual Care — Participants in the usual care (UC) group met in-person once a month with either a pharmacist or dietician for the duration of the 6-month intervention. The focus of these sessions was on facilitating the adoption and maintenance of health behaviors related to diet, physical activity and sleep to promote weight loss. These participants were set up on the Nudge app, but they did not use the mHWC (texting) feature.
  Arms: Usual Care

SUMMARY:
The objective of this study was to assess the effectiveness of a 6-month text-based mobile health and wellness (mHWC) intervention, as compared to usual care (UC), for weight loss in adults. Participants were randomly assigned to one of the two groups (mHWC or UC). At the beginning of the study, both groups were given a Fitbit wearable device, and a weight scale. All participants also received a counseling session from a dietician focused on diet, physical activity, and sleep, and were set up on the Nudge app, a commercially-available mHWC platform. Participants in the mHWC group received text-based coaching messages via Nudge and did not return to the clinic for the duration of the 6-month intervention. Those in the UC group met once a month with a pharmacist or dietician for 6 months. In both groups, the focus was on facilitating health behavior change related to diet, physical activity, and sleep to promote weight loss.

We hypothesized that weight loss at 6 months would be greater in the mHWC group vs. the UC group.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27 kg/m^2
* Waist circumference ≥35 inches (women) or ≥40 inches (men)
* Own an Android smartphone or iPhone capable of running the Nudge and Fitbit applications.
* Indicate sending at least one text-based (e.g., SMS, Facebook, Twitter) message via their smartphone on most days

Exclusion Criteria:

* Pregnant
* Pacemaker or other electronic implant
* Weight ≥400 pounds
* Weight loss ≥5% of bodyweight in previous 6 months
* High cardiovascular risk, as determined by Physical Activity Readiness Questionnaire (PAR-Q) and physician review, as needed.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 6 months (mean 193 ± 21 days)
  Assessed at baseline and follow-up

SECONDARY OUTCOMES:
Change Waist Circumference | 6 months (mean 193 ± 21 days)
  Assessed at baseline and follow-up
Change in Self-Reported Physical Activity | 6 months (mean 193 ± 21 days)
  Assessed via Exercise Vital Sign (EVS) at baseline and follow-up. The EVS is used to assess via self-report the amount of physical activity or exercise an individual engages in during an average week. It asks: 1. On average, how many days a week do you perform physical activity or exercise, such as walking or jogging? and 2. On average, how many minutes of physical activity or exercise do you perform on those days?
Change in Self-Reported Sleep Quantity | 6 months (mean 193 ± 21 days)
  Assessed via Pittsburgh Sleep Quality Index (PSQI) at baseline and follow-up. The PSQI is used to assess via self-report an individual's nightly average sleep quality and quantity over the previous 30 day period. As for quality, the higher the score, the lower the quality of sleep.
Change in Self-Reported Daily Caloric Consumption | 6 months (mean 193 ± 21 days)
  Assessed via the Automated Self-Assessment 24-hour (ASA24) Dietary Assessment at baseline and follow-up. The ASA24 is a detailed 24-hour food recall that can be used to estimate via self-report diet quality and quantity.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Hollingsworth, PharmD, PhD, Principal Investigator — VCOM-Auburn
Locations (1):
- Auburn University Pharmaceutical Care Center, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share IPD with other researchers.